CLINICAL TRIAL: NCT06753695
Title: Prevalence of Hypomineralized Second Primary Molars(HSPM) and Its Association with Dental Hypersensitivity in a Group of Egyptian Children: a Cross-sectional Study.
Brief Title: Prevalence of Hypomineralized Second Primary Molars and Their Association with Dental Hypersensitivity in Egyptian Children
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mamdouh Ibrahim, Dentist and Principal Investigato, Cairo University
Other Study IDs: HSPM-DH-EG-2024
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hypomineralized Second Primary Molars; Dental Hypersensitivity
Keywords: HSPM; DH; hypo-mineralized second primary molars; hypomineralized E

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
hypomineralized second primary molars and dental hypersensitivity in a group of Egyptian children

DETAILED DESCRIPTION:
the prevalence of the condition of hypomineralized second primary molars in a group of Egyptian children and the association of this condition to dental hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children
* cooperative patients both genders and included 4-9 years old children at least one HSPM affected molar and one non affected molar absence of syndromes or craniofacial anomalies

Exclusion Criteria:

* other developmental defects(amelogensis imperfecta ...) children ongoing anti-inflammatory drugs children who caregiver will not sign the informed consent

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: a group of gentian children aged form4 to 9 years old
Sampling Method: Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
EAPD scoring criteria and wurzberg scroring system | 1 year
  present/absent of the condition

SECONDARY OUTCOMES:
VAS scale and SCASS scale | 1year
  measuring dental hypersensitivity using VAS scale and SCASS scale to reach for an association of dental hypersensitivity and HSPM

CONTACTS AND LOCATIONS:
Overall Officials: Aya M Ibrahim, B.D.S., Principal Investigator — University of Cairo, Department of Dentistry.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD will be available within 12 months following publication of the primary results.